CLINICAL TRIAL: NCT00388661
Title: Double Blind Placebo-controlled Study on the Efficacy of Melatonin on Sleep, Resulting in an Improved Quality of Life in Hemodialysis Patients
Brief Title: Melatonin and Quality of Life in Dialysis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meander Medical Center (Other)
Collaborators: Dutch Kidney Foundation (Other)
Responsible Party: Department of Clinical Pharmacy, Meander Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-06.31 M / Melody; R-06.31 M
Record Dates: First submitted 2006-10-16; First posted 2006-10-17 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Sleep Problems; Haemodialysis
Keywords: sleep problems; quality of life; melatonin; sleep apnea; medication; preload; nutritional status; ProBNP
MeSH Terms: conditions — Parasomnias; Sleep Apnea Syndromes | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Melatonin (Active Comparator): melatonin 3mg
  Interventions: Drug: Melatonin tablet 3 mg once daily
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: Melatonin tablet 3 mg once daily — Melatonin tablet 3 mg once daily
  Arms: Melatonin
Drug: Placebo comparator — Placebo comparator
  Arms: Placebo

SUMMARY:
Sleep problems can lead to a bad quality of life and a raise of morbidity, also in dialysis patients. Sleep problems can be caused by a disturbance of circadian rhythms in our body. For a good regulation of these circadian rhythms a uniform external synchronisation is necessary. This is the synchronisation of the biological clock of our body by light and other influences. In case of a disturbance of the external synchronisation, due to for example naps during the day or wake periods at night, internal rhythms can be unlinked. As a result a weakened melatonin rhythm and a problematic sleep-wake cycle can be observed. Most dialysis patients have sleep problems. Their sleep latency is prolonged. They often take a nap during the day and their sleep efficiency is poor. There has only been one study on the melatonin rhythm of dialysis patients. The conclusion of this study was that the melatonin rhythm of dialysis patients is weakened and disturbed, probably caused by renal insufficiency. In this study no link was made between melatonin rhythm and the nature and severity of possible sleep problems. In different studies with non-dialysis patients and a disturbed melatonin rhythm, exogenous melatonin at the right time leads to a recovery of the normal rhythm and the normal biological clock and a better quality of life.

The aim is to improve quality of life of hemodialysis patients with a placebo-controlled study with melatonin to investigate if exogenous melatonin can improve sleep problems and on the longer term improve quality of life (and secondary morbidity) of dialysis patients.

DETAILED DESCRIPTION:
Objective of the study:

Does melatonin by improving sleep parameters improve quality of life of hemodialysis patients?

Study design:

Placebo-controlled, double-blind, randomized trial

Study population:

hemodialysis patients

Intervention:

melatonin 3 mg once daily (or placebo)

Primary study parameters/outcome of the study:

1. improvement of vitality (dimension quality of life) by 15 points (RAND SF 36)
2. improvement general health by 15 points (dimension quality of life, RAND SF 36)

Secondary study parameters/outcome of the study:

1. Change in biochemical parameters
2. Change in ProBNP
3. Change in nutritional status
4. Change in use of medication
5. Change in preload

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* Man/Women between 18 and 85 years
* Understanding and knowledge of the dutch language
* End Stage Renal Disease, stable chronic hemodialysis > 3 months
* SpKt/V(total) > 1,2 pro dialysis
* Validated actometer shows that sleep efficiency < 90% or sleep latency > 15 minutes or fragmentation index > 25 points

Exclusion Criteria:

* Known major illness, which interferes with patient's participation in the study according to the investigator)or which results in a probable patient's survival of less than 1 year.
* Instable angina pectoris, heart failure NYHA class IV
* Pregnancy
* Current use of melatonin of known allergy of melatonin
* Participation in other medication/drug research within a month before inclusion

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2007-04; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Improvement of vitality (dimension quality of life) by 15 points (RAND SF 36) | 6-12 months
Improvement general health by 15 points (dimension quality of life, RAND SF 36) | 6-12 months

SECONDARY OUTCOMES:
Change in biochemical parameters | 3-6-9-12 months
Change in ProBNP | 12 months
Change in nutritional status | 12 months
Change in use of medication | 6-12 months
Change in preload | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pieter ter Wee, MD, PhD, Study Chair — Amsterdam UMC, location VUmc
Locations (2):
- Netherlands (2):
  - Meander Medical Center, Amersfoort
  - Kennemer Gasthuis, Haarlem